CLINICAL TRIAL: NCT00043602
Title: Clinician Managed Interpersonal Psychotherapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Scott Stuart, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH059668 (NIH); R01MH059668 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2002-08-09; First posted 2002-08-13 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Depression; Depression, Postpartum
MeSH Terms: conditions — Depression; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive clinician-managed interpersonal psychotherapy
  Interventions: Behavioral: Clinician managed interpersonal psychotherapy (CM-IPT)
- 2 (Active Comparator): Participants will receive standard interpersonal psychotherapy
  Interventions: Behavioral: Standard interpersonal psychotherapy (IPT)

INTERVENTIONS:
Behavioral: Standard interpersonal psychotherapy (IPT) — Participants will receive 12 sessions of IPT over 12 weeks.
  Arms: 2
Behavioral: Clinician managed interpersonal psychotherapy (CM-IPT) — Participants will receive 12 sessions of CM-IPT over 1 year.
  Arms: 1

SUMMARY:
This 12-week study will evaluate the effectiveness of Clinician-Managed Interpersonal Psychotherapy (CM-IPT) in treating postpartum depression and will compare CM-IPT to standard IPT.

DETAILED DESCRIPTION:
CM-IPT is delivered in 12 sessions over the course of a year. Standard IPT is delivered in 12 sessions in the first 12 weeks after treatment assignment.

ELIGIBILITY:
Inclusion criteria:

* Women between 8 and 24 weeks postpartum
* Meet DSM-IV criteria for Major Depression
* Hamilton Rating Scale for Depression score of 12 or more

Exclusion criteria:

* Active substance abuse
* Psychotic disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2001-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | Measured at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Scott P. Stuart, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States